CLINICAL TRIAL: NCT06352294
Title: The Effects of Myofascial Relaxation Technique Applied Together With Core Stabilization Trainings on Balance, Pain, Joint Range of Motion and Functionality in Individuals With Chronic Neck Pain
Brief Title: Examining The Effects of Core Stabilization Exercises and Myofascial Release Technique in Individuals With Chronic Neck Pain: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Muhammed Samed DALAKÇI, Lecturer, Kirsehir Ahi Evran Universitesi
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MSDALAKCI
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Neck Pain
Keywords: Balance; Functionality; Myofascial relase
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Core stability training (Active Comparator): A total of 18 sessions of core stabilization training will be given to the participants in 6 weeks.
  Interventions: Other: Core stability training
- Basic stability training and myofascial relasing method (Experimental): Core stabilization training and myfacial relaxation application will be performed to the participants for 6 weeks and 18 sessions.
  Interventions: Other: Core stability training and myofascial relase

INTERVENTIONS:
Other: Core stability training — Before starting core stabilization exercises, hotpack will be given for 15 minutes in the warm-up phase, TENS application, then craniocervical flexion training will be given. Core stabilization exercises consist of three stages: easy, medium and difficult
  Arms: Core stability training
Other: Core stability training and myofascial relase — Before starting core stabilization exercises, hotpack will be given for 15 minutes in the warm-up phase, TENS application, then craniocervical flexion training will be given. Core stabilization exercises consist of three stages: easy, medium and difficult. In addition, myofascial relaxation will be applied with roller bar along the superficial back line.
  Arms: Basic stability training and myofascial relasing method

SUMMARY:
Chronic neck pain is a musculoskeletal disorder that affects people frequently in life.

Postural control is based on the process of correctly identifying and selectively focusing the incoming afferent input of the Central Nervous System (CNS).

The main treatment options for people with neck pain include soft tissue and joint mobilizations, stabilization exercises for the neck, trunk and shoulder muscles, cervical Deckings, relaxation training, strengthening exercises and body awareness and posture training.

In this study, it was aimed to investigate the effects of myofascial relaxation on balance, pain, joint range of motion and functionality in individuals with chronic neck pain by dividing them into two groups in the form of core stabilization and core stabilization and myofascial relaxation.

The study included 45 people between the ages of 18 and 65. In two groups, the core stabilization group will be 22 people, and the core stabilization and myofascial relaxation group will be 23 people. The study period is planned as 6 weeks and 3 sessions per week.

ELIGIBILITY:
Inclusion Criteria:

* Having neck pain that has been going on for at least three months
* The mean pain intensity according to the Visual Analog Scale (GAS) is moderate [4-6.9 centimeters (cm)
* December] or be at a severe (7 cm and above) level
* To be between the ages of Dec 18-65
* To be literate and to be a writer
* Volunteering to participate in the study

Exclusion Criteria:

* Having severe degenerative arthritis
* Having a neurological finding due to spinal root compression (Positive upper limb stretching tests,cervical compression test)
* To have a finding due to pressure of the spinal cord (Positive L'hermitte sign, Babinski sign) is
* Having undergone cervical spine surgery
* Having a cervical neck fracture and/or joint subluxation/dislocation
* Having osteoporosis and/or neck pain due to a tumor
* Having a history of primary malignancy
* Being pregnant
* The title refers to neurological disease (Parkinson's, Multiple Sclerosis, etc.)
* Having received physiotherapy and rehabilitation in the last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-06-14 (Actual); Study Completion 2024-06-14 (Actual)

PRIMARY OUTCOMES:
Pain severity | 6 weeks
  Visual Analog Scale ( 0-10, higher means worse )
Pressure pain threshold (PPT) | 6 weeks
  Pressure pain threshold was measured with an algometer.

SECONDARY OUTCOMES:
Balance | 6 weeks
  Measurements were made with a Biodex balance device. The scores obtained as a result of 3 measurements were averaged. As the score increases, the balance is considered to have worsened.
Range of motion | 6 weeks
  Movement skills of the neck area were recorded.
Neck Disability İndex | 6 weeks
  It is a disability level determination scale consisting of 10 questions for the person with neck pain.
DASH | 6 weeks
  It is a 30-question survey used to determine the level of functionality in patients suffering from upper extremity and neck pain. As the score increases, the level of disability increases.

CONTACTS AND LOCATIONS:
Locations (1):
- Kırşehir Ahi Evran Üniversitesi, Merkez, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No